CLINICAL TRIAL: NCT01418703
Title: Feasibility Study of a Modular Control to Range System in T1DM
Brief Title: Feasibility Study of a Modular Control to Range System in Type 1 Diabetes Mellitus
Acronym: MDB003
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Virginia (Other)
Collaborators: Abbott Diabetes Care (Industry); Insulet Corporation (Industry); DexCom, Inc. (Industry); University of California, Santa Barbara (Other)
Responsible Party: Principal Investigator, Marc Breton, Associate Professor, University of Virginia
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Supportive Care
Other Study IDs: 14356
Record Dates: First submitted 2011-07-08; First posted 2011-08-17 (Estimated); Results first posted 2014-11-13 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Type 1 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 1

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Closed Loop Control (CLC) (Experimental): The CLC used a computer to make recommendations for their insulin treatment. This study arm was designed to demonstrate management of glucose using a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). This system was designed to both:
  * monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  * predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Interventions: Device: Closed Loop Control (CLC)
- Open Loop (Placebo Comparator): The subject were in charge of their insulin treatment.
  Interventions: Device: Open Loop

INTERVENTIONS:
Device: Closed Loop Control (CLC) — In this study, the researchers compared the management of diabetes during physical activity and meals with the closed-loop system developed at the University of Virginia. This Control to Range System uses two DexCom Seven Continuous Glucose Monitor, a computer containing an investigational control algorithm (well-defined instructions that are expressed in mathematical equations), and an OmniPod Insulin Management System, a portable subcutaneous (under the skin) insulin pump. During the closed-loop admission, the computer used CGM values to make recommendations of insulin treatment based on the algorithms.
  Arms: Closed Loop Control (CLC)
Device: Open Loop — This admission was to assess the subjects' level of glucose control and created a base to compare the performance of the closed-loop system. Subjects monitored their own blood glucose values and administer their basal/bolus as they would at home. Subjects use their own pump. Otherwise, the admission remained the same as in the closed-loop admission (i.e. meals, exercise, etc...).
  Arms: Open Loop

SUMMARY:
In this protocol the investigators plan to demonstrate the feasibility of a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). The protocol is designed to challenge the insulin management system with meals and mild exercise, so as to demonstrate its capacity to avoid large glucose excursion with changing metabolic state. This system is designed to both

* monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
* predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.

The investigators plan to enroll 12 adult Type 1 Diabetes Mellitus (T1DM) patients (expected retention 10/12) and compare glucose control performances under two treatments: standard vs. the new insulin management system. The protocol will include a total of 6 admissions per subject (4 out-patients and 2 in-patients): screening, effort test, CGM insertion 1, inpatient 1, CGM insertion 2, and inpatient 2. During the 24h inpatient admissions, the patients will be challenged with 30 minutes of mild exercise and 3 meals, insulin coverage of these events will vary depending on the chosen treatment, each subject will be exposed to both studied treatments (repeated measure design).The order of treatment during the inpatient admissions will be randomized.

ELIGIBILITY:
Inclusion Criteria:

* 21 years of age and up to and including 65 years of age.
* Have Type 1 Diabetes Mellitus as defined by American Diabetes Association criteria or judgment of physician for at least 2 years (including those who may also be treated with metformin, thiazolidinedione, exenatide, or pramlintide).
* Use of an insulin pump
* If on antihypertensive, thyroid, anti-depressant or lipid lowering medication, have stability on the medication for at least 2 months prior to enrollment in the study
* Willingness to use lispro (Humalog) insulin for the duration of the inpatient study
* Demonstration of proper mental status and cognition for the study
* Willingness to stop using any dietary supplements for two weeks prior to admission and for the duration of their participation.

Exclusion Criteria:

* Age <21or >65
* Pregnancy
* Hematocrit <36% (females); <38% (males)
* HemoglobinA1c > 10.0
* Symptomatic coronary artery disease (e.g. history of myocardial infarction, history of acute coronary syndrome, history of therapeutic coronary intervention, history of coronary bypass or stenting procedure, stable or unstable angina, episode of chest pain of cardiac etiology with documented EKG changes, positive stress test or catheterization with coronary blockages >50%).
* Use of a medication that significantly lowers heart rate (beta blockers, reserpine, guanethidine, methyldopa, clonidine, cimetidine, digitalis, calcium channel blockers, amiodarone, antiarrythmic drugs, or lithium)
* Congestive heart failure
* History of a cerebrovascular event
* Use of a medication that significantly impacts glucose metabolism (oral steroids)
* Atrial fibrillation
* Uncontrolled hypertension (resting blood pressure >140/90)
* History of a systemic or deep tissue infection with methicillin- resistant staph aureus or Candida albicans
* Use of a device that may pose electromagnetic compatibility issues and/or radiofrequency interference with the FreeStyle NavigatorTM CGM (implantable cardioverter-defibrillator, electronic pacemaker, neurostimulator,intrathecal pump, and cochlear implants)
* Active enrollment in another clinical trial
* Allergy or adverse reaction to lispro insulin
* Known adrenal gland problem, pancreatic tumor, or insulinoma
* Current alcohol abuse by patient history, substance abuse by patient history, or severe mental illness
* Retinopathy and renal failure
* Uncontrolled anxiety or panic disorder
* Known bleeding diathesis or dyscrasia
* Renal insufficiency (creatinine >1.5)
* Any comorbid condition affecting glucose metabolism

Ages: 21 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2009-10; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marc D Breton, Ph.D., Principal Investigator — University of Virgnia - School of Medicine, Psychiatry and Neurobehavioral Sciences
Locations (1):
- University of Virginia Health System, Charlottesville, Virginia, United States

REFERENCES:
- [Result] Breton M, Farret A, Bruttomesso D, Anderson S, Magni L, Patek S, Dalla Man C, Place J, Demartini S, Del Favero S, Toffanin C, Hughes-Karvetski C, Dassau E, Zisser H, Doyle FJ 3rd, De Nicolao G, Avogaro A, Cobelli C, Renard E, Kovatchev B; International Artificial Pancreas Study Group. Fully integrated artificial pancreas in type 1 diabetes: modular closed-loop glucose control maintains near normoglycemia. Diabetes. 2012 Sep;61(9):2230-7. doi: 10.2337/db11-1445. Epub 2012 Jun 11. PMID 22688340

RESULTS

PARTICIPANT FLOW:
Groups:
- Open-Loop First, Then sCTR Closed-Loop: Completed open-loop, then sCTR (Standard Control to Range ) Closed-Loop admission.
  The two modules of sCTR are the SSM (safety supervision module) and a standard range control module that avoids prolonged hyperglycemic excursions. Both modules use a real-time estimate of the patient 's metabolic state based on CGM (continuous glucose monitor) and insulin infusion data. This estimate is used for prediction of the risks of hypo-and hyperglycemia 30-45 min ahead of the event. If a risk for hypoglycemia is predicted, the SSM attenuates automatically any insulin requests proportionally to the predicted risk level. How aggressively the system attenuates insulin is determined with patient characteristics (e.g. body weight, insulin-to-carbohydrate ratio, and basal insulin delivery). If a risk for hyperglycemia is predicted, the range controller gives a correction bolus using the predicted plasma glucose and the patient's CSII (continuous subcutaneous insulin infusion) parameters.
- sCTR Closed-Loop First, Then Open-Loop: Participants completed sCTR Closed-Loop admission, then completed open-loop admission.
  The two modules of sCTR are the SSM and a standard range control module that avoids prolonged hyperglycemic excursions. Both modules use a real-time estimate of the patient 's metabolic state based on CGM and insulin infusion data. This estimate is used for prediction of the risks of hypo-and hyperglycemia 30-45 min ahead of the event. If a risk for hypoglycemia is predicted, the SSM attenuates automatically any insulin requests proportionally to the predicted risk level. How aggressively the system attenuates insulin is determined with patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery). If a risk for hyperglycemia is predicted, the range controller gives a correction bolus using the predicted plasma glucose and the patient's CSII parameters; the system injects only half of the computed bolus and can do so once every hour.
- Open-Loop First, Then eCTR Closed-Loop: Participants completed open-loop admission, then completed eCTR (Enhanced Control to Range) closed-loop admission.
  The two modules of the eCTR are the SSM and an enhanced range control module based on an MPC (model predictive control) algorithm that aims to maintain glycemia in a target range. eCTR also uses insulin-on-board constraints (29) intended to prevent insulin overdose during intensified therapy. The rationale behind MPC was presented in detail in a recent review (7). Controller aggressiveness was individualized for each subject based on readily available patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery) (30). In this application, the MPC worked using information from the individual's conventional therapy. Premeal boluses were triggered by the patient, with the carbohydrate amount measured in the clinical research center (CRC) kitchen but automatically calculated by eCTR.
- eCTR Closed-Loop First, Then Open-Loop: Participants completed open-loop admission, then completed eCTR closed-loop admission.
  The two modules of the eCTR are the SSM and an enhanced range control module based on an MPC algorithm that aims to maintain glycemia in a target range. eCTR also uses insulin-on-board constraints (29) intended to prevent insulin overdose during intensified therapy. The rationale behind MPC was presented in detail in a recent review (7). Controller aggressiveness was individualized for each subject based on readily available patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery) (30). In this application, the MPC worked using information from the individual's conventional therapy. Premeal boluses were triggered by the patient, with the carbohydrate amount measured in the CRC kitchen but automatically calculated by eCTR.
Period: Overall Study
Arm/Group | Open-Loop First, Then sCTR Closed-Loop | sCTR Closed-Loop First, Then Open-Loop | Open-Loop First, Then eCTR Closed-Loop | eCTR Closed-Loop First, Then Open-Loop
Started | 13 | 13 | 6 | 6
Completed | 13 | 13 | 6 | 6
Not Completed | 0 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Standard Control to Range (sCTR): The two modules of sCTR are the SSM and a standard range control module that avoids prolonged hyperglycemic excursions. Both modules use a real-time estimate of the patient 's metabolic state based on CGM and insulin infusion data. This estimate is used for prediction of the risks of hypo-and hyperglycemia 30-45 min ahead of the event. If a risk for hypoglycemia is predicted, the SSM attenuates automatically any insulin requests proportionally to the predicted risk level. How aggressively the system attenuates insulin is determined with patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery). If a risk for hyperglycemia is predicted, the range controller gives a correction bolus using the predicted plasma glucose and the patient's CSII parameters; the system injects only half of the computed bolus and can do so once every hour.
- Enhanced Control to Range (eCTR): The two modules of the eCTR are the SSM and an enhanced range control module based on an MPC algorithm that aims to maintain glycemia in a target range. eCTR also uses insulin-on-board constraints (29) intended to prevent insulin overdose during intensified therapy. The rationale behind MPC was presented in detail in a recent review (7). Controller aggressiveness was individualized for each subject based on readily available patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery) (30). In this application, the MPC worked using information from the individual's conventional therapy. Premeal boluses were triggered by the patient, with the carbohydrate amount measured in the CRC kitchen but automatically calculated by eCTR.
- Total: Total of all reporting groups
Arm/Group | Standard Control to Range (sCTR) | Enhanced Control to Range (eCTR) | Total
Number analyzed (Participants) | 26 | 12 | 38
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 11 | 0 | 11
  Between 18 and 65 years | 15 | 12 | 27
  >=65 years | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 11 | 4 | 15
  Male | 15 | 8 | 23

OUTCOME MEASURES:

1. Primary Outcome: Hypoglycemic Events
Description: Number of hypoglycemic events below 70 mg/dL per patient per day
Time Frame: Throughout each 22-hour closed-loop and open-loop admission for sCTR and eCTR
Measure: Mean (Standard Deviation); unit: events/admission per patient
Groups:
- Closed Loop: The CLC used a computer to make recommendations for their insulin treatment. This study arm was designed to demonstrate management of glucose using a modular insulin management system based on continuous glucose monitoring and targeted towards the avoidance of hypoglycemic and prolonged hyperglycemic episodes (i.e. control to range). This system was designed to both:
  * monitor the meal boluses of the patient and correct it in case of observed/predicted under insulinization (avoidance of prolonged hyperglycemia), based on a coarse and subjective knowledge of the meal amount, a precise understanding of the subject's day to day insulin treatment, continuous glucose monitoring, and past insulin injections;
  * predict and avoid hypoglycemic events, based on continuous glucose reading and past insulin injection.
  Closed Loop Control (CLC): During the closed-loop admission, the computer used CGM values to make recommendations of insulin treatment based on the algorithms.
Arm/Group | Open Loop | Closed Loop
Number analyzed (Participants) | 38 | 38
events/admission per patient
  sCTR (N=26) | 1.08 (0.27) | 0.4 (0.13)
  eCTR (N=12) | 1.4 (0.56) | 1.6 (0.68)

2. Secondary Outcome: Percent Time Spent in Near Normoglycemia
Description: Comparison of time spent in near normoglycemia (3.9 to 10 mmol/mL) in open-loop vs closed-loop sCTR and eCTR.
Time Frame: Throughout each 22-hour closed-loop and open-loop admission for sCTR and eCTR
Measure: Mean (Standard Deviation); unit: percentage of time
Arm/Group | Open Loop | Closed Loop
Number analyzed (Participants) | 38 | 38
percentage of time
  sCTR (N=26) | 61.5 (5.2) | 74.4 (3.9)
  eCTR (N=12) | 76.8 (5.0) | 90.1 (3.4)

3. Secondary Outcome: Mean Glucose
Description: Average plasma glucose concentration in mg/dl
Time Frame: Throughout each 22-hour closed-loop and open-loop admission for sCTR and eCTR
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Open Loop | Closed Loop
Number analyzed (Participants) | 38 | 38
mg/dL
  sCTR (N=26) | 8.82 (0.54) | 8.34 (0.28)
  eCTR (N=12) | 7.74 (0.44) | 6.68 (0.28)

ADVERSE EVENTS:
Groups:
- Open-Loop: This admission was to assess the subjects' level of glucose control and created a base to compare the performance of the closed-loop system. Subjects monitored their own blood glucose values and administer their basal/bolus as they would at home. Subjects use their own pump. Otherwise, the admission remained the same as in the closed-loop admission (i.e. meals, exercise, etc...).
- sCTR Closed-Loop Control: The two modules of sCTR are the SSM and a standard range control module that avoids prolonged hyperglycemic excursions. Both modules use a real-time estimate of the patient 's metabolic state based on CGM and insulin infusion data. This estimate is used for prediction of the risks of hypo-and hyperglycemia 30-45 min ahead of the event. If a risk for hypoglycemia is predicted, the SSM attenuates automatically any insulin requests proportionally to the predicted risk level. How aggressively the system attenuates insulin is determined with patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery). If a risk for hyperglycemia is predicted, the range controller gives a correction bolus using the predicted plasma glucose and the patient's CSII parameters; the system injects only half of the computed bolus and can do so once every hour.
- eCTR Closed-Loop Control: The two modules of the eCTR are the SSM and an enhanced range control module based on an MPC algorithm that aims to maintain glycemia in a target range. eCTR also uses insulin-on-board constraints (29) intended to prevent insulin overdose during intensified therapy. The rationale behind MPC was presented in detail in a recent review (7). Controller aggressiveness was individualized for each subject based on readily available patient characteristics (e.g., body weight, insulin-to-carbohydrate ratio, and basal insulin delivery) (30). In this application, the MPC worked using information from the individual's conventional therapy. Premeal boluses were triggered by the patient, with the carbohydrate amount measured in the CRC kitchen but automatically calculated by eCTR.
Arm/Group | Open-Loop | sCTR Closed-Loop Control | eCTR Closed-Loop Control
Serious Adverse Events (participants affected / at risk) | 0/38 | 0/26 | 0/12
Other Adverse Events (participants affected / at risk) | 2/38 | 2/26 | 0/12
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Open-Loop (N=38) | sCTR Closed-Loop Control (N=26) | eCTR Closed-Loop Control (N=12)
Hyperglycemia (Endocrine disorders) | 0 (0) | 2 (2) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0)
Vasovagal Episode (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes